CLINICAL TRIAL: NCT01493739
Title: EBUS-TBNA for Diagnosis of Mediastinal Lymphadenopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHIH-HSI KUO, Principle Investigator, Consultant Physician, Respiratory Medicine Department, Chang Gung Memorial Hospital
Other Study IDs: EBUSTBNA_01
Record Dates: First submitted 2011-11-21; First posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Mediastinal Lymphadenopathy; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lymphadenopathy

SUMMARY:
This study aims on the combinatorial results of cytology, histopathology and microbiology obatined by EBUS-TBNA for unselected mediastina lesions.

DETAILED DESCRIPTION:
A number of studies have proved EBUS-TBNA to be useful for lymph node staging in lung cancer. The diagnostic performance is equivalent to mediastinoscopy while the invasiveness is far less. This study primarily focusing on merged approach of cytology, histopathology and microbioloogy obatined by EBUS-TBNA for unselected mediastina lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* mediastinal lymphadenopathy on Chest CT scan
* with a short-axis > 10mm

Exclusion Criteria:

* patients intolerant to bronchoscopy exam
* unstable vital sign (Blood pressure, heart rate, breath rate)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mediastinal lymphadenopathy on Chest CT scan with a short-axis > 10mm
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate | Participant will be followed within an average of three months

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hso Kuo, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taipei, Taiwan